CLINICAL TRIAL: NCT01751243
Title: Transplantation of Hematopoietic Progenitors From Haploidentical Donor With Selective in Vitro Depletion Allo-reactive Lymphocytes in Patient With High Risk Hematological Malignancies.
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Andalusian Initiative for Advanced Therapies - Fundación Pública Andaluza Progreso y Salud (Other)
Collaborators: Iniciativa Andaluza en Terapias Avanzadas (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALODEPLETE
Record Dates: First submitted 2012-12-13; First posted 2012-12-17 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2017-09

CONDITIONS: Transplant-Related Hematologic Malignancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group 0 (Placebo Comparator): Haploidentical transplantation of hematopoietic progenitors
  Interventions: Other: Haploidentical transplantation of hematopoietic progenitors
- Group 1 (Experimental): Allo-depleted lymphocyte infusion dose: 1x105 CD3/Kg
  Interventions: Other: Allo-depleted lymphocyte infusion
- Group 2 (Experimental): Allo-depleted lymphocyte infusion dose: 3x105 CD3/Kg
  Interventions: Other: Allo-depleted lymphocyte infusion
- Group 3 (Experimental): Allo-depleted lymphocyte infusion dose: 5x105 CD3/Kg
  Interventions: Other: Allo-depleted lymphocyte infusion
- Group 4 (Experimental): Allo-depleted lymphocyte infusion dose: 1x106 CD3/Kg
  Interventions: Other: Allo-depleted lymphocyte infusion
- Group 5 (Experimental): Allo-depleted lymphocyte infusion dose: 3x106 CD3/Kg
  Interventions: Other: Allo-depleted lymphocyte infusion

INTERVENTIONS:
Other: Allo-depleted lymphocyte infusion — Doses: 1x105 CD3/Kg; 3x105 CD3/Kg; 5x105 CD3/Kg; 1x106 CD3/Kg;31x106 CD3/Kg;
  Arms: Group 1; Group 2; Group 3; Group 4; Group 5
Other: Haploidentical transplantation of hematopoietic progenitors — Haploidentical transplantation of hematopoietic progenitors without subsequent infusion of allo-depleted lymphocytes.
  Arms: Group 0

SUMMARY:
Therapeutic exploratory study to evaluate safety, open, nonrandomized, multicentre, prospective, of cohort of patients who will receive different doses of allo-depleted lymphocytes .

This project joins in this pioneering worldwide initiative with its own technology based on the use of proteasome inhibitors in vitro, which advantages are, over other methods described, the continuing viability of regulatory T cells and the use of a product to generate allo-depletion that, contrary to those reported by other research groups, it does not pose problems from the point of view of its use or toxicity as we employ a drug widely used clinically by intravenous administration.

DETAILED DESCRIPTION:
The main objective of the study is to determine the safety of transplantation of hematopoietic progenitors from haploidentical donor with in vitro allo-depleted lymphocyte infusion.

Secondary objectives:

* To assess the immune reconstitution pre and post-infusion of allo-depleted lymphocytes.
* To analyze the incidence of infections (CMV and aspergillus) post-transplant.
* To analyze the impact of acute and chronic graft-versus-host disease (GVHD).
* To optimize the dose of allo-depleted lymphocytes to reconstitute an immune response against pathogens without causing GVHD.
* To assess the rate of graft and myeloid and platelet engraftment time.
* To assess the rate of relapses, event-free survival and overall survival. It is hoped to recruit 20 clinically evaluable patients for safety purpose.

The inclusion period is not more than 2 ½ years. Study duration shall not exceed three years from the inclusion of the first patient. The minimum follow-up of patients is 6 months after transplantation.

The first 5 patients (group 0) will receive haploidentical transplantation of hematopoietic progenitors without subsequent infusion of allo-depleted lymphocytes and then in cohorts of 3 patients, infuse +4 post-transplant day at doses of: 1x105 cluster of differentiation 3 (CD3)/kg(group 1), 3x105 CD3/kg (group 2), 5x105 CD3 / kg (group 3), 1x106 CD3/kg (group 4) and 3x106 CD3/kg (group 5).

Donor: it is performed one leukapheresis at least 30 days (4 weeks) prior to the scheduled progenitors infusion (day 0), in order to obtain effector T cells.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged between 16 and 50 years.
* Diagnosed as Hematological malignancy candidates to allogeneic transplant lacking of related or unrelated suitable donor (is more than one Human leukocyte antigen (HLA) mismatched over 8 antigens) and who don't have a cord with an adequate cellularity. The minimum period of search to be able to include the patient in the trial, currently considering the medium to find a suitable donor to be 2 months, it is set to 10 weeks, although in specific situations in which the responsible physician considers that the patient has a high risk of relapse, it may be proceed with inclusion before that period. These cases will be assessed individually with the trial coordinator.

Exclusion Criteria:

* General condition> Eastern Cooperative Oncology Group (ECOG) scale 2.
* Left Ventricular ejection fraction (LVEF) <39%.
* Diffusion capacity of lung for carbon monoxide (DLCO) and forced vital capacity (FVC) <39% of the theoretical values.
* Impaired liver function (total bilirubin higher than 2 mg / dL and / or transaminases higher than 3 times the normal maximum.
* Creatinine clearance <50 mL / minute.
* Presence of symptomatic heart, liver cirrhosis or chronic active hepatitis.
* Active tuberculosis.
* Serious diseases which prevent chemotherapy treatments.
* Associated neoplasias (active neoplasias which, according to the opinion of the investigator and the sponsor, could jeopardize patient safety).
* Presence of associated psychiatric pathology.
* HIV infection.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events and serious adverse events after allo-depleted lymphocyte infusion in vitro. | 6 months

SECONDARY OUTCOMES:
Incidence of acute and chronic GVHD | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jose-Antonio Perez-Simón, MD, PhD, Principal Investigator — University Hospital Virgen del Rocío; Antonio Torres, MD, PhD, Principal Investigator — University Hospital Reina Sofía; Lucía Lopez-Corral, MD, PhD, Principal Investigator — University Hospital de Salamanca; Mª Ángeles Cuesta, MD, PhD, Principal Investigator — University Hospital Carlos Haya
Locations (4):
- Spain (4):
  - University Hospital Reina Sofia, Córdoba
  - University Hospital Carlos Haya, Málaga
  - University Hospital de Salamanca, Salamanca
  - University Hospital Virgen del Rocío, Seville

REFERENCES:
- See also: Andalusian Molecular Biology and Regenerative Medicine Centre — http://www.cabimer.es